CLINICAL TRIAL: NCT04952467
Title: An Open Label, Single-dose, Single-period Study to Assess the Pharmacokinetics, Mass Balance Recovery, Metabolite Profile and Metabolite Identification of 14C-XEN1101 in Healthy Male Subjects
Brief Title: Single-dose Mass Balance Recovery and Metabolite Profile and Identification of 14C-XEN1101
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xenon Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: XPF-008-103; 2021-000735-32 (EudraCT Number)
Record Dates: First submitted 2021-06-27; First posted 2021-07-07 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Healthy Volunteers
Keywords: XEN1101; Mass Balance; Phase 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Drug: (14C)-XEN1101 (Experimental): Subjects will receive oral 14C-XEN1101 under fed conditions.
  Interventions: Drug: 14C-XEN1101

INTERVENTIONS:
Drug: 14C-XEN1101 — Subjects will receive a single oral administration of a capsule containing 20 mg XEN1101

SUMMARY:
This study will evaluate the mass balance recovery and metabolite profile, and will identify metabolite structures following a single oral dose of 14C-XEN1101 in healthy adult male subjects.

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) of 18.0 to 32.0 kg/m2
* Must be willing and able to communicate and participate in the whole study
* Provide written informed consent
* Adhere to the specified contraception requirements

Key Exclusion Criteria:

* Subjects who have received any investigational medicinal product (IMP) in a clinical research study within 90 days
* Evidence of any current infection or an infection within 14 days before study drug administration
* History of any drug or alcohol abuse in the past 2 years
* Subjects with pregnant or lactating partners
* Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 millisievert (mSv) in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 2017, shall participate in the study
* Participation in a clinical trial involving administration of radiolabelled compound(s) within 180 days of the planned dosing date of this study
* Clinically significant abnormal clinical chemistry, haematology, coagulation or urinalysis. Subjects with Gilbert's Syndrome will be excluded.
* Confirmed positive drugs of abuse test result
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) antibody results
* History of clinically significant cardiovascular, renal, hepatic, dermatological, chronic respiratory or gastrointestinal disease, neurological or psychiatric disorder
* Donation of blood or plasma within the previous 3 months or loss of greater than 400 mL of blood

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2021-10-04 (Actual); Study Completion 2021-10-04 (Actual)

PRIMARY OUTCOMES:
Total radioactivity excreted in urine and faeces following oral administration of XEN1101 | From Screening up to Day 57 post-dose
  Cumulative amount of total radioactivity excreted in urine and feces combined (CumAe(total)) and expressed as a % of the radioactive dose administered (Cum%Ae(total)) following oral administration of 14C-XEN1101

SECONDARY OUTCOMES:
14C Metabolite profiling in of plasma, urine and feces | From Screening up to Day 57 post-dose
  Chemical structure of each metabolite classified as >10% (by AUC) of total radioactivity in plasma and >10% dose excreted in urine and faeces following oral administration of XEN1101
Pharmacokinetic (PK) data for 14C-XEN1101; Tmax | From Screening up to Day 57 post-dose
  Time of maximum observed concentration for XEN1101 and metabolites in plasma and for total radioactivity in plasma and whole blood following oral administration of 14C-XEN1101
PK data for 14C-XEN1101; Cmax | From Screening up to Day 57 post-dose
  Maximum observed concentration for XEN1101 and metabolites in plasma and for total radioactivity in plasma and whole blood following oral administration of 14C-XEN1101
PK data for 14C-XEN1101; T1/2 | From Screening up to Day 57 post-dose
  Terminal elimination half-life for XEN1101 and metabolites in plasma and for total radioactivity in plasma and whole blood following oral administration of 14C-XEN1101
Mass balance data for 14C-XEN1101 in urine | From Screening up to Day 57 post-dose
  CumAe(urine)expressed as a percentage of the radioactive dose administered (Cum%Ae(urine))
Mass balance data for 14C-XEN1101 in feces | From Screening up to Day 57 post-dose
  CumAe(feces) expressed as a percentage of the radioactive dose administered Cum%Ae(feces)
Plasma whole blood concentration ratios for total radioactivity | From Screening up to Day 57 post-dose
  Evaluation of whole blood:plasma concentration ratios for total radioactivity for corresponding time points
Frequency and severity of treatment-emergent adverse events (TEAEs), treatment-emergent serious adverse events (SAEs), and TEAEs leading to treatment discontinuations | From Screening up to Day 57 post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Xenon Pharmaceuticals Inc.
Locations (1):
- Quotient Sciences, Ruddington, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No